CLINICAL TRIAL: NCT00003652
Title: Intensification Therapy for Locally Advanced Epidermoid Cancer of the Anal Canal - Phase III Intergroup Study
Brief Title: Combination Chemotherapy Plus Radiation Therapy in Treating Patients With Stage II or Stage III Anal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066744; FNCLCC-FFCD-SFRO-ACCORD-3; EU-98050
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Anal Cancer
Keywords: stage II anal cancer; stage III anal cancer; squamous cell carcinoma of the anus; cloacogenic carcinoma of the anus; basaloid carcinoma of the anus
MeSH Terms: conditions — Anus Neoplasms; Anal Canal Carcinoma | interventions — Cisplatin; Fluorouracil; Neoadjuvant Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: cisplatin
Drug: fluorouracil
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy with radiation therapy may kill more tumor cells.

PURPOSE: This randomized phase III trial is studying different regimens of giving combination chemotherapy together with radiation therapy and comparing how well they work in treating patients with stage II or stage III anal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of concurrent chemotherapy and radiotherapy with or without neoadjuvant chemotherapy with fluorouracil and cisplatin in patients with stage II or III anal canal cancer.
* Compare the efficacy of two levels of radiation dose in patients with stage II or III anal canal cancer.
* Compare the sphincter conservation of the anus by these regimens.
* Compare the effect of these regimens on survival and quality of life of these patients.

OUTLINE: This is a randomized, multicenter study.

Patients are randomized to one of four treatment arms.

* Arm I: Patients receive induction chemotherapy consisting of fluorouracil IV over 24 hours on days 1-4 and cisplatin IV over 1 hour on day 1 or 2 every 4 weeks for 2 courses. Beginning 4 weeks later, patients receive chemoradiotherapy. This regimen consists of fluorouracil IV over 24 hours on days 1-4 and cisplatin IV over 1 hour on day 1 or 2 and repeated 4 weeks later, plus pelvic radiotherapy beginning on day 1 and continuing for 5 weeks (once a day, 5 days/week). Patients receive low dose radiotherapy directly to the tumor beginning 3 weeks later and continuing for 2 weeks.
* Arm II: Patients receive induction chemotherapy and chemoradiotherapy as in arm I, plus high dose radiotherapy directly to the tumor.
* Arm III (control arm): Patients receive chemoradiotherapy and low dose radiotherapy to the tumor as in arm I.
* Arm IV: Patients receive chemoradiotherapy and high dose radiotherapy to the tumor as in arm II.

After study treatment is completed, patients with nonfixed inguinal tumors may undergo surgical resection followed by radiotherapy or radiotherapy alone. Patients with fixed inguinal tumors may receive further radiotherapy alone.

Quality of life is assessed before treatment, at 2 months after completion of treatment, and at 5 years.

Patients are followed every 4 months for 2 years, every 6 months for 3 years, then annually thereafter.

PROJECTED ACCRUAL: A total of 350 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven nonmetastatic anal cancer

  * Anal/rectal junction OR
  * Anal/cutaneous junction with the majority of the tumor in the anal canal, above the junction
  * Epidermoid cancer (well-differentiated, fairly differentiated, or basaloid) OR
  * Cloacogenic cancer
  * Stage II or III

    * T2 at least 4 cm OR
    * T3 OR
    * T4, N0-3, M0 OR
    * T1, N1-3 OR
    * T2 (less than 4 cm), N1-3
* Tumors at least 4 cm in greatest dimension and/or tumors with lymph node invasion must be nonmetastatic by ultrasound
* No prior surgery to remove tumor

PATIENT CHARACTERISTICS:

Age:

* 80 and under

Performance status:

* WHO 0 or 1

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 2,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 11 g/dL (transfusion allowed)

Hepatic:

* Not specified

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* No cardiac condition contraindicating use of fluorouracil

Other:

* No prior malignancy within 5 years except squamous cell or basal cell skin cancer or carcinoma in situ of the cervix or breast
* No other serious medical or psychological condition
* No serious immunosuppression

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior biologic therapy

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* No prior endocrine therapy

Radiotherapy:

* No prior pelvic or inguinal radiotherapy

Surgery:

* See Disease Characteristics
* No prior definitive colostomy

Ages: 0 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 1999-01-04 (Actual); Primary Completion 2006-04-01 (Actual); Study Completion 2007-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Didier Peiffert, MD, Study Chair — Centre Alexis Vautrin
Locations (48):
- France (48):
  - Centre Paul Papin, Angers
  - Institut Sainte Catherine, Avignon
  - Institut Bergonie, Bordeaux
  - CHU Ambroise Pare, Boulogne-Billancourt
  - C.H. Bourg En Bresse, Bourg-en-Bresse
  - Centre Regional Francois Baclesse, Caen
  - Centre Hospitalier, Chalon-sur-Saône
  - Hopital Louis Pasteur, Colmar
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon
  - Centre Hospitalier Departemental, La Roche-sur-Yon
  - Centre Oscar Lambret, Lille
  - Centre Hospital Regional Universitaire de Limoges, Limoges
  - Centre Leon Berard, Lyon
  - Institut J. Paoli and I. Calmettes, Marseille
  - CHU de la Timone, Marseille
  - Hopital Clinique Claude Bernard, Metz
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Centre Hospitalier de Mulhouse, Mulhouse
  - Centre D'Oncologie De Gentilly, Nancy
  - Centre Catherine de Sienne, Nantes
  - Centre Regional Rene Gauducheau, Nantes-Saint Herblain
  - Centre Antoine Lacassagne, Nice
  - CHR D'Orleans - Hopital de la Source, Orléans
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Bichat - Claude Bernard, Paris
  - Hopital Robert Debre, Paris
  - Institut Curie - Section Medicale, Paris
  - Hopital Saint-Louis, Paris
  - CHU Pitie-Salpetriere, Paris
  - Hopital Tenon, Paris
  - Hopital Jean Bernard, Poitiers
  - Clinique Ste - Marie, Pontoise
  - Institut Jean Godinot, Reims
  - Centre Eugene Marquis, Rennes
  - Hopital Charles Nicolle, Rouen
  - Centre Henri Becquerel, Rouen
  - Clinique Armoricaine De Radiologie, Saint-Brieuc
  - Centre Rene Huguenin, Saint-Cloud
  - Centre Hospitalier General de Saint Nazaire, Saint-Nazaire
  - Clinique de l'Orangerie, Strasbourg
  - Centre Paul Strauss, Strasbourg
  - Centre Hospitalier Regional Metz Thionville, Thionville
  - Institut Claudius Regaud, Toulouse
  - Clinique Fleming, Tours
  - Nouvelle Clinique Generale, Valence
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Result] Tournier-Rangeard L, Mercier M, Peiffert D, Gerard JP, Romestaing P, Lemanski C, Mirabel X, Pommier P, Denis B. Radiochemotherapy of locally advanced anal canal carcinoma: prospective assessment of early impact on the quality of life (randomized trial ACCORD 03). Radiother Oncol. 2008 Jun;87(3):391-7. doi: 10.1016/j.radonc.2007.12.004. Epub 2008 Jan 11. PMID 18191265